CLINICAL TRIAL: NCT00545688
Title: A Randomized, Open Label Study to Compare the Complete Pathological Response Rate Achieved With 4 Combinations of Herceptin, Docetaxel and Pertuzumab in Patients With Locally Advanced, Inflammatory or Early Stage HER2 Positive Breast Cancer
Brief Title: A Study of Pertuzumab in Combination With Herceptin in Patients With HER2 Positive Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO20697
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel; pertuzumab

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Herceptin; Drug: Docetaxel
- 2 (Experimental)
  Interventions: Drug: Herceptin; Drug: Docetaxel; Drug: Pertuzumab
- 3 (Experimental)
  Interventions: Drug: Herceptin; Drug: Pertuzumab
- 4 (Experimental)
  Interventions: Drug: Docetaxel; Drug: Pertuzumab

INTERVENTIONS:
Drug: Herceptin — 8mg/kg iv loading dose, followed by 6mg/kg iv 3-weekly
  Other Names: Trastuzumab
  Arms: 1; 2; 3
Drug: Docetaxel — 75mg/m2 iv escalating to 100mg/m2 iv 3-weekly
  Arms: 1; 2; 4
Drug: Pertuzumab — 840mg iv loading dose, followed by 420mg iv 3-weekly
  Arms: 2; 3; 4

SUMMARY:
This 4 arm study will evaluate the efficacy and safety of 4 neoadjuvant treatment regimens in female patients with locally advanced, inflammatory or early stage HER2 positive breast cancer. Before surgery, patients will be randomized to one of 4 treatment arms, to receive 4 cycles of a)Herceptin + docetaxel b)Herceptin + docetaxel + pertuzumab c)Herceptin + pertuzumab or 4)pertuzumab + docetaxel. Pertuzumab will be administered at a loading dose of 840mg iv, then 420mg iv 3-weekly, Herceptin at a loading dose of 8mg/kg iv then 6mg/kg 3-weekly, and docetaxel at a dose of 75mg/m2 escalating to 100mg/m2 3-weekly. During the entire pre- and post-surgery period all patients will receive adequate chemotherapy as per standard of care, as well as any surgery and/or radiotherapy as required. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=18 years of age;
* locally advanced, inflammatory or early stage invasive breast cancer;
* HER2 positive (HER2+++ by IHC or FISH/CISH+).

Exclusion Criteria:

* metastatic disease (Stage IV) or bilateral breast cancer;
* previous anticancer therapy or radiotherapy for any malignancy;
* other malignancy, other than cancer in situ of the cervix, or basal cell cancer;
* insulin-dependent diabetes;
* clinically relevant cardiovascular disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2006-06-26 (Actual); Primary Completion 2014-09-22 (Actual); Study Completion 2014-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (77):
- Australia (2):
  - Geelong Hospital; Andrew Love Cancer Centre, Geelong, Victoria
  - Mount Medical Center, Perth, Western Australia
- Austria (2):
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I, Vienna
  - Kaiser Franz Josef Spital; Iii. Medizinische Abt. Mit Onkologie, Vienna
- Brazil (9):
  - Hospital de Caridade de Ijui; Oncologia, Ijuí, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Faculdade de Medicina do ABC - FMABC; Oncologia e Hematologia, Santo André, São Paulo
  - Instituto do Cancer Arnaldo Vieira de Carvalho - ICAVC; Pesquisa Clinica, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Inst. Brasileiro de Controle Ao Cancer; Oncologia Clinica / Quimioterapia, São Paulo, São Paulo
  - Instituto de Oncologia de Sorocaba - CEPOS, Sorocaba, São Paulo
- Canada (5):
  - Moncton Hospital, Moncton, New Brunswick
  - Cancer Centre of Southeastern Ontario; Kingston General Hospital, Kingston, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - McGill University; Montreal General Hosptial; Oncology, Montreal, Quebec
  - CHU de Québec - Hôpital du Saint-Sacrement / ONCOLOGY, Québec
- Israel (3):
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Meir Medical Center; Oncology, Kfar Saba
  - Sourasky / Ichilov Hospital; Dept. of Oncology, Tel Aviv
- Italy (9):
  - Az. Osp. S. Orsola Malpighi; Istituto Di Oncologia Seragnoli, Bologna, Emilia-Romagna
  - Ospedale Regionale Di Parma; Divisione Di Oncologia Medica, Parma, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria Dipartimento Interaziendale Di Oncologia, Udine, Friuli Venezia Giulia
  - ASST OVEST MILANESE; Oncologia Medica, Legnano, Lombardy
  - Ospedale San Raffaele, Servizio di Oncologia e Chemioterapia, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 1, Milan, Lombardy
  - Ospedale Calvi di Noale; U.O. Complessa di Oncologia ed Ematologia Oncologica, Mirano, Veneto
  - Polo Ospedaliero Santorso, Santorso, Veneto
  - Ospedale Di Vicenza; Nefrologia, Oncologia Medica, Vicenza, Veneto
- Mexico (3):
  - Hospital Miguel Hidalgo, Aguascalientes
  - ARKE Estudios Clínicos S.A. de C.V., Mexico City
  - Issstep Puebla, ; Oncology, Puebla City
- Peru (2):
  - Instituto Regional de Enfermedades Neoplásicas del Sur; Centro de Inv. de Medicina Oncológica, Arequipa
  - Hospital Nacional Edgardo Rebagliati Martins; Oncologia, Lima
- Poland (7):
  - Samodzielny Publiczny Kliniczny Nr 1 W Lublinie; Klinika Chirurgii Onkologicznej, Lublin
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Olsztyński Ośrodek Onkologiczny Kopernik sp. z o.o., Olsztyn
  - Oddzial Chemioterapii Szpitala Klinicznego Nr 1 w Poznaniu, Poznan
  - NZOZ Centrum Medyczne HCP Sp. z o.o., Poznan
  - Central Hospital of Military School of Medicine; Oncology, Warsaw
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
- Russia (11):
  - FSBI "Scientific Research Institute of Oncology named after N.N.Petrov" Ministry of Health of RF, Saint Petersburg, Sankt-Peterburg
  - SI of Healthcare Kazan Oncology Dispensary, Kazan'
  - Russian Oncology Research Center n.a. N.N. Blokhin Dpt of Clinical Pharmacology and Chemotherapy, Moscow
  - NSI of Healthcare Central Clinical Hospital #2 n.a. N.A.Semashko of the Russian Railways, Moscow
  - State Institution Of Healthcare Republican Oncology Dispensary, Petrozavodsk
  - State Budget Institution of Healthcare of Stavropol region Pyatigorsk Oncology Dispensary, Pyatigorsk
  - SBI for HPE "Ryazan State Medical University n.a. I.P. Pavlov" of MoH of RF, Ryazan
  - SBI of Healthcare Leningrad Regional Oncology Dispensary, Saint Petersburg
  - SBI of Healthcare Samara Regional Clinical Oncology Dispensary, Samara
  - SI of HealthCare Oncologic Dispensary #2 of department of healthcare of Krasnodar region, Sashi
  - Ulyanovsk Regional Oncology Dispensary; Chemotherapy, Ulyanovsk
- South Korea (2):
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
- Spain (8):
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital de Cruces; Servicio de Oncologia, Barakaldo, Vizcaya
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (2):
  - Karolinska Hospital; Oncology - Radiumhemmet, Stockholm
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Switzerland (2):
  - Kantonsspital Baden; Frauenklinik, Baden
  - Brustzentrum, Zurich
- Taiwan (3):
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
- Thailand (3):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Prince of Songkla Uni ; Unit of Medical Oncology, Songkhla
- Turkey (Türkiye) (2):
  - Dokuz Eylul Uni Medical Faculty; Oncology Dept, Izmir
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sıhhiye, Ankara
- United Kingdom (2):
  - Walsgrave Hospital; Dept of Oncology, Coventry
  - Christie Hospital; Breast Cancer Research Office, Manchester

REFERENCES:
- [Derived] Bianchini G, Kiermaier A, Bianchi GV, Im YH, Pienkowski T, Liu MC, Tseng LM, Dowsett M, Zabaglo L, Kirk S, Szado T, Eng-Wong J, Amler LC, Valagussa P, Gianni L. Biomarker analysis of the NeoSphere study: pertuzumab, trastuzumab, and docetaxel versus trastuzumab plus docetaxel, pertuzumab plus trastuzumab, or pertuzumab plus docetaxel for the neoadjuvant treatment of HER2-positive breast cancer. Breast Cancer Res. 2017 Feb 9;19(1):16. doi: 10.1186/s13058-017-0806-9. PMID 28183321
- [Derived] Swain SM, Schneeweiss A, Gianni L, Gao JJ, Stein A, Waldron-Lynch M, Heeson S, Beattie MS, Yoo B, Cortes J, Baselga J. Incidence and management of diarrhea in patients with HER2-positive breast cancer treated with pertuzumab. Ann Oncol. 2017 Apr 1;28(4):761-768. doi: 10.1093/annonc/mdw695. PMID 28057664
- [Derived] Gianni L, Pienkowski T, Im YH, Tseng LM, Liu MC, Lluch A, Staroslawska E, de la Haba-Rodriguez J, Im SA, Pedrini JL, Poirier B, Morandi P, Semiglazov V, Srimuninnimit V, Bianchi GV, Magazzu D, McNally V, Douthwaite H, Ross G, Valagussa P. 5-year analysis of neoadjuvant pertuzumab and trastuzumab in patients with locally advanced, inflammatory, or early-stage HER2-positive breast cancer (NeoSphere): a multicentre, open-label, phase 2 randomised trial. Lancet Oncol. 2016 Jun;17(6):791-800. doi: 10.1016/S1470-2045(16)00163-7. Epub 2016 May 11. PMID 27179402
- [Derived] Gianni L, Pienkowski T, Im YH, Roman L, Tseng LM, Liu MC, Lluch A, Staroslawska E, de la Haba-Rodriguez J, Im SA, Pedrini JL, Poirier B, Morandi P, Semiglazov V, Srimuninnimit V, Bianchi G, Szado T, Ratnayake J, Ross G, Valagussa P. Efficacy and safety of neoadjuvant pertuzumab and trastuzumab in women with locally advanced, inflammatory, or early HER2-positive breast cancer (NeoSphere): a randomised multicentre, open-label, phase 2 trial. Lancet Oncol. 2012 Jan;13(1):25-32. doi: 10.1016/S1470-2045(11)70336-9. Epub 2011 Dec 6. PMID 22153890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 107, 107, 107, and 96 participants (total 417) were randomized to Arms Trastuzumab plus (+) Docetaxel (T+ D) , Trastuzumab+Pertuzumab+Docetaxel (T+Ptz+D), Trastuzumab+Pertuzumab (T+Ptz), and Pertuzumab+Docetaxel (Ptz+D), respectively and were included in intent-to-treat population (as randomized).
Pre-assignment Details: 3 participants did not receive correct treatment, as randomized, and 1 (in Arm Trastuzumab + Docetaxel) did not receive any treatment. Safety population (as treated) included 107, 107, 108, and 94 participants in Arms 'T+D', 'T+Ptz+D', 'T+Ptz', and 'Ptz+D', respectively. Participant flow was available for "As Treated" participants.
Groups:
- Trastuzumab + Docetaxel: Neoadjuvant (Pre-Operative) Treatment: Participants received trastuzumab intravenous (IV) infusion at a loading dose of 8 milligrams per kilogram (mg/kg) on Day 1 of Cycle 1 (21-day cycle) followed by a maintenance dose of 6 mg/kg on Day 1 of Cycles 2-4 and docetaxel IV infusion at a starting dose of 75 milligrams per square meter (mg/m^2) on Day 1 of Cycle 1 followed by 100 mg/m^2 on Day 1 of Cycles 2-4, if no dose limiting toxicity occurred.
  Adjuvant (2-Week Post-Operative) Treatment: Participants received trastuzumab 6 mg/kg IV followed by 5-fluorouracil 600 mg/m^2 IV, epirubicin 90 mg/m^2 IV, and cyclophosphamide 600 mg/m^2 IV (FEC) on Day 1 and every 3 weeks thereafter for three cycles (Cycles 5-7). Trastuzumab 6 mg/kg IV was continued every 3 weeks from Cycle 8 to Cycle 17.
- Trastuzumab+Pertuzumab+Docetaxel: Neoadjuvant (Pre-Operative) Treatment: Participants received trastuzumab IV infusion at a loading dose of 8 mg/kg and pertuzumab IV infusion at a loading dose of 840 mg on Day 1 of Cycle 1 (21-day cycle) followed by a maintenance dose of 6 mg/kg trastuzumab and 420 mg pertuzumab on Day 1 of Cycles 2-4. Docetaxel IV infusion was administered at a starting dose of 75 mg/m^2 on Day 1 of Cycle 1 followed by 100 mg/m^2 on Day 1 of Cycles 2-4, if no dose limiting toxicity occurred.
  Adjuvant (2-Week Post-Operative) Treatment: Participants received trastuzumab 6 mg/kg IV followed by FEC on Day 1 and every 3 weeks thereafter for three cycles (Cycles 5-7). Trastuzumab 6 mg/kg IV was continued every 3 weeks from Cycle 8 to Cycle 17.
- Trastuzumab+Pertuzumab: Neoadjuvant (Pre-Operative) Treatment: Participants received trastuzumab IV infusion at a loading dose of 8 mg/kg and pertuzumab IV infusion at a loading dose of 840 mg on Day 1 of Cycle 1 (21-day cycle) followed by a maintenance dose of 6 mg/kg trastuzumab and 420 mg pertuzumab on Day 1 of Cycles 2-4.
  Adjuvant (2-Week Post-Operative) Treatment: Participants received trastuzumab 6 mg/kg IV followed by docetaxel 75 mg/m^2 IV on Day 1 of Cycle 5 followed by docetaxel 100 mg/m^2 for three cycles (Cycles 6-8) if no dose-limiting toxicity occurred. For Cycles 9 to 11, participants received trastuzumab 6 mg/kg IV followed by FEC on Day 1 and every 3 weeks thereafter for three cycles. Trastuzumab 6 mg/kg IV was continued every 3 weeks from Cycle 12 until Cycle 17.
- Pertuzumab+Docetaxel: Neoadjuvant (Pre-Operative) Treatment: Participants received pertuzumab IV at a loading dose of 840 mg on Day 1 of Cycle 1 (21-day cycle) followed by a maintenance dose of 420 mg on Day 1 of Cycles 2-4. Docetaxel IV infusion was administered at a starting dose of 75 mg/m^2 on Day 1 of Cycle 1 followed by 100 mg/m^2 on Day 1 of Cycles 2-4, if no dose limiting toxicity occurred.
  Adjuvant (2-Week Post-Operative) Treatment: Participants received trastuzumab 6 mg/kg IV followed by FEC on Day 1 and every 3 weeks thereafter for three cycles (Cycles 5-7). Trastuzumab 6 mg/kg IV was continued every 3 weeks from Cycle 8 to Cycle 21.
Period: Neo-Adjuvant Treatment Period
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Started | 107 | 107 | 108 | 94
Completed | 103 | 102 | 94 | 88
Not Completed | 4 | 5 | 14 | 6
Not completed — Protocol Violation | 1 | 2 | 1 | 1
Not completed — Refused Treatment | 1 | 1 | 4 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 7 | 2
Not completed — Unknown Reason | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 2
Period: Adjuvant Treatment Period
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Started | 103 | 102 | 94 | 88
Completed | 98 | 94 | 90 | 74
Not Completed | 5 | 8 | 4 | 14
Not completed — Disease Progression | 3 | 3 | 0 | 7
Not completed — Refused Treatment | 1 | 1 | 1 | 5
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 3 | 2 | 2
Not completed — Unknown Reason | 0 | 1 | 0 | 0
Period: Follow-Up Period
Arm/Group | Trastuzumab + Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Started | 98 | 102 | 98 | 87
Completed | 77 | 83 | 78 | 60
Not Completed | 21 | 19 | 20 | 27
Not completed — Death | 4 | 2 | 2 | 6
Not completed — Disease Progression | 6 | 5 | 9 | 9
Not completed — Refused Treatment | 6 | 2 | 0 | 2
Not completed — Lost to Follow-up | 3 | 3 | 3 | 1
Not completed — Unspecified Reason | 2 | 5 | 6 | 8
Not completed — Violation of Selection Criteria at Entry | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) Population included all randomized participants who received any amount of study medication. Analysis was performed according to initial randomization.
Groups:
- Trastuzumab+Docetaxel: Neoadjuvant (Pre-Operative) Treatment: Participants received trastuzumab IV infusion at a loading dose of 8 mg/kg on Day 1 of Cycle 1 (21-day cycle) followed by a maintenance dose of 6 mg/kg on Day 1 of Cycles 2-4 and docetaxel IV infusion at a starting dose of 75 mg/m^2 on Day 1 of Cycle 1 followed by 100 mg/m^2 on Day 1 of Cycles 2-4, if no dose limiting toxicity occurred.
  Adjuvant (2-Week Post-Operative) Treatment: Participants received trastuzumab 6 mg/kg IV followed by FEC on Day 1 and every 3 weeks thereafter for three cycles (Cycles 5-7). Trastuzumab 6 mg/kg IV was continued every 3 weeks from Cycle 8 to Cycle 17.
- Total: Total of all reporting groups
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel | Total
Number analyzed (Participants) | 107 | 107 | 107 | 96 | 417
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (8.94) | 49.6 (10.05) | 49.7 (10.67) | 48.9 (10.50) | 49.8 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 107 | 107 | 96 | 417
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Pathological Complete Response (pCR)
Description: pCR was defined as an absence of invasive neoplastic cells at microscopic examination of the tumor remnants after surgery following primary systemic therapy. Participants with invalid/missing pCR assessments were defined as non-responders
Time Frame: Approximately 4 months from randomization following surgery or early withdrawal, whichever occurred first (Surgery was performed within 2 weeks after Cycle 4)
Population: ITT Population; Analysis was performed according to initial randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 107 | 107 | 107 | 96
percentage of participants | 29.0 [20.6 to 38.5] | 45.8 [36.1 to 55.7] | 16.8 [10.3 to 25.3] | 24.0 [15.8 to 33.7]
Statistical Analysis 1: Comparison: Trastuzumab+Docetaxel vs Trastuzumab+Pertuzumab+Docetaxel; Test type: Superiority or Other; p = 0.0094, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test stratified by breast cancer type (operable, locally advanced, or inflammatory) and estrogen and or progesterone positivity (either positive versus both negative); Difference in Response rates = 16.82, 95% CI 2-sided [3.5 to 30.1]
Statistical Analysis 2: Comparison: Trastuzumab+Docetaxel vs Trastuzumab+Pertuzumab+Docetaxel; Test type: Superiority or Other; p = 0.0141, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test, with Simes multiplicity adjustment
Statistical Analysis 3: Comparison: Trastuzumab+Docetaxel vs Trastuzumab+Pertuzumab; Test type: Superiority or Other; p = 0.0198, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Response rates = -12.15, 95% CI 2-sided [-23.8 to -0.5]
Statistical Analysis 4: Comparison: Trastuzumab+Docetaxel vs Trastuzumab+Pertuzumab; Test type: Superiority or Other; p = 0.0198, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test, with Simes multiplicity adjustment
Statistical Analysis 5: Comparison: Trastuzumab+Pertuzumab+Docetaxel vs Pertuzumab+Docetaxel; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Difference in Response rates = -21.84, 95% CI 2-sided [-35.1 to -8.5]
Statistical Analysis 6: Comparison: Trastuzumab+Pertuzumab+Docetaxel vs Pertuzumab+Docetaxel; Test type: Superiority or Other; p = 0.0030, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test, with Simes multiplicity adjustment

2. Secondary Outcome: Percentage of Participants Achieving Best Primary Tumor Response (Complete Response [CR], Partial Response [PR], Stable Disease [SD] or Disease Progression [PD]) During Neo-Adjuvant Treatment by X-Ray/Mammography
Description: Tumor assessments were made based upon the Response Evaluation Criteria in Solid Tumors (RECIST) criteria - version 1.0. The clinical response at each cycle up to the last assessment prior to surgery was derived for primary breast tumor using the following algorithm: CR: if measurement of '0' is noted at a given cycle as compared to baseline measurement which is greater than (>)0 at screening or cycle 1 Day 1; PR: if measurement is at least a 30 percent (%) decreased compared to baseline levels . (Reference= baseline size or sum of sizes); SD: if measurement at a given cycle is not sufficient shrinkage to qualify for neither PR nor sufficient increase to qualify for PD compared to baseline levels. PD: if lesion is at least a 20 % increase from measurements at baseline.
Time Frame: Baseline up to Cycle 4 (assessed at, Baseline and Day 1 of Cycles 1-4 Pre-Surgery) Up to approximately 24 months
Population: ITT Population; Analysis was performed according to initial randomization. Number of participants analyzed = participants evaluable for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 71 | 58 | 61 | 47
percentage of participants
  CR | 18.3 | 19.0 | 13.1 | 19.1
  PR | 49.3 | 46.6 | 36.1 | 46.8
  SD | 31.0 | 32.8 | 44.3 | 34.0
  PD | 1.4 | 1.7 | 6.6 | 0.0

3. Primary Outcome: Percentage of Participants Achieving pCR by Breast Cancer Type
Description: pCR was defined as an absence of invasive neoplastic cells at microscopic examination of the tumor remnants after surgery following primary systemic therapy. Based on the type of breast cancer participants were categorized as those with 1. Operable breast cancer, 2. Inflammatory breast cancer and 3. Locally advanced breast cancer. Participants with invalid/missing pCR assessments were defined as non-responders.
Time Frame: as for outcome 1
Population: ITT Population; Analysis was performed according to initial randomization. Number (n) equal (=) number of participants included in the specified type of breast cancer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 107 | 107 | 107 | 96
percentage of participants
  Operable Breast Cancer (n=64,65,65,60) | 23.4 [13.8 to 35.7] | 47.7 [35.1 to 60.5] | 16.9 [8.8 to 28.3] | 26.7 [16.1 to 39.7]
  Inflammatory Breast Cancer (n=7,10,7,5) | 14.3 [0.4 to 57.9] | 40.0 [12.2 to 73.8] | 28.6 [3.7 to 71.0] | 40.0 [5.3 to 85.3]
  Locally Advance Breast Cancer (36,32,35,31) | 41.7 [25.5 to 59.2] | 43.8 [26.4 to 62.3] | 14.3 [4.8 to 30.3] | 16.1 [5.5 to 33.7]

4. Primary Outcome: Percentage of Participants Achieving pCR by Hormone Receptor Status
Description: pCR was defined as an absence of invasive neoplastic cells at microscopic examination of the tumor remnants after surgery following primary systemic therapy. Participants were classified as Estrogen and/or Progesterone positive (+ve), Estrogen and/or Progesterone negative (-ve) or receptor status unknown. Participants with invalid/missing pCR assessments were defined as non-responders.
Time Frame: as for outcome 1
Population: ITT Population; Analysis was performed according to initial randomization. n = number of participants included in the specified hormone receptor status.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 107 | 107 | 107 | 96
percentage of participants
  Estrogen and/or Progesterone +ve (n=50,50,51,46) | 20.0 [10.0 to 33.7] | 26.0 [14.6 to 40.3] | 5.9 [1.2 to 16.2] | 17.4 [7.8 to 31.4]
  Estrogen and/or Progesterone -ve (n=57,57,55,50) | 36.8 [24.4 to 50.7] | 63.2 [49.3 to 75.6] | 27.3 [16.1 to 41.0] | 30.0 [17.9 to 44.6]
  Receptor Status Unknown (0,0,1,0) | NA [NA to NA] — There were no participants in this category. | NA [NA to NA] — There were no participants in this category. | 0.0 [0.0 to 97.5] | NA [NA to NA] — There were no participants in this category.

5. Primary Outcome: Percentage of Participants Achieving pCR by Lymph Node Status
Description: pCR was defined as an absence of invasive neoplastic cells at microscopic examination of the tumor remnants after surgery following primary systemic therapy. Lymph node status was defined as either negative lymph node at surgery or positive lymph node at surgery. Participants with invalid/missing pCR assessments were defined as non-responders.
Time Frame: as for outcome 1
Population: ITT Population; Analysis was performed according to initial randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 107 | 107 | 107 | 96
percentage of participants
  pCR achieved and Negative Lymph Nodes at Surgery | 21.5 | 39.3 | 11.2 | 17.7
  pCR achieved and Positive Lymph Nodes at Surgery | 7.5 | 6.5 | 5.6 | 6.3

6. Primary Outcome: Percentage of Participants Achieving pCR by Presence or Absence of Residual Intraductal Carcinoma (DCIS) / Intalobular Carcinoma (LCIS)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: ITT Population; Analysis was performed according to initial randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 107 | 107 | 107 | 96
percentage of participants
  pCR Achieved and No residual DCIS/LCIS at Surgery | 16.8 | 36.4 | 9.3 | 17.7
  pCR Achieved and Residual DCIS/LCIS at Surgery | 12.1 | 9.3 | 7.5 | 6.3

7. Secondary Outcome: Percentage of Participants Achieving Best Overall Response (CR, PR, SD or PD) During Neo-Adjuvant Period by X-Ray/Mammography
Description: Tumor assessments were made based on the RECIST criteria - version 1.0 The overall response at each cycle up to the last assessment prior to surgery was derived for: i) the primary breast lesion; (ii) across secondary breast lesions, (iii) across all breast lesions (iv) across axillary nodes (v) across supraclavicular nodes and (vi) across all nodes (vii) across all lesions (overall) using the following algorithm: CR: if measurement of '0' is noted at a given cycle as compared to baseline measurement which is >0 at screening or cycle 1 day 1; PR: if measurement is at least a 30% decreased compared to baseline levels . (Reference= baseline size or sum of sizes); SD: if measurement at a given cycle is not sufficient shrinkage to qualify for neither PR nor sufficient increase to qualify for PD compared to baseline levels. PD: if lesion is at least a 20 % increase from measurements at baseline. Overall response is derived based on the sum total of breast tumors and all nodes examined.
Time Frame: Baseline up to Cycle 4 (assessed at Baseline, Day 1 of Cycles 1-4 Pre-Surgery) Up to approximately 24 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 71 | 53 | 55 | 43
percentage of participants
  CR | 18.3 | 18.9 | 12.7 | 18.6
  PR | 49.3 | 49.1 | 34.5 | 46.5
  SD | 31.0 | 30.2 | 45.5 | 34.9
  PD | 1.4 | 1.9 | 7.3 | 0.0

8. Secondary Outcome: Percentage of Participants Achieving Best Primary Breast Tumor Response (CR, PR, SD or PD) During Neo-Adjuvant Period by Clinical Examination
Description: Tumor assessments were made based on the RECIST criteria - version 1.0 The clinical response at each cycle up to the last assessment prior to surgery was derived for primary breast tumor using the following algorithm: CR: if measurement of '0' is noted at a given cycle as compared to baseline measurement which is >0 at screening or cycle 1 day 1; PR: if measurement is at least a 30% decreased compared to baseline levels . (Reference= baseline size or sum of sizes); SD: if measurement at a given cycle is not sufficient shrinkage to qualify for neither PR nor sufficient increase to qualify for PD compared to baseline levels. PD: if lesion is at least a 20 % increase from measurements at baseline. Overall response is derived based on the sum total of breast tumors and all nodes examined.
Time Frame: Baseline up to Cycle 4 (assessed at Baseline, Day 1 of Cycles 1-4 Pre-Surgery) Up to approximately 24 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 99 | 101 | 102 | 91
percentage of participants
  CR | 23.2 | 30.7 | 16.7 | 20.9
  PR | 56.6 | 57.4 | 51.0 | 50.5
  SD | 20.2 | 11.9 | 30.4 | 28.6
  PD | 0.0 | 0.0 | 2.0 | 0.0

9. Secondary Outcome: Percentage of Participants Achieving Best Overall Response (CR, PR, SD or PD) During the Neo-Adjuvant Period by Clinical Examination
Description: Tumor assessments were made based on the RECIST criteria - version 1.0 The clinical response at each cycle up to the last assessment prior to surgery was derived for: i) the primary breast lesion; (ii) across secondary breast lesions, (iii) across all breast lesions (iv) across axillary nodes (v) across supraclavicular nodes and (vi) across all nodes (vii) across all lesions (overall) using the following algorithm: CR: if measurement of '0' is noted at a given cycle as compared to baseline measurement which is >0 at screening or cycle 1 day 1; PR: if measurement is at least a 30% decreased compared to baseline levels . (Reference= baseline size or sum of sizes); SD: if measurement at a given cycle is not sufficient shrinkage to qualify for neither PR nor sufficient increase to qualify for PD compared to baseline levels. PD: if lesion is at least a 20 % increase from measurements at baseline. Overall response is derived based on the sum total of breast tumors and all nodes examined.
Time Frame: Baseline up to Cycle 4 (assessed at Baseline, Day 1 of Cycles 1-4 Pre-Surgery) Up to approximately 24 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 97 | 100 | 98 | 88
percentage of participants
  CR | 21.6 | 25.0 | 11.2 | 15.9
  PR | 59.8 | 63.0 | 55.1 | 58.0
  SD | 17.5 | 12.0 | 31.6 | 26.1
  PD | 1.0 | 0.0 | 2.0 | 0.0

10. Secondary Outcome: Percentage of Participants Achieving Clinical Response During Neo-Adjuvant Period by X-Ray/Mammography
Description: Clinical response was determined based on tumor measurements by sponsor in combination with tumor response assessment by investigator. Tumor assessments were made based on the RECIST criteria - version 1.0 The clinical response at each cycle up to the last assessment prior to surgery was derived for: i) the primary breast lesion; (ii) across secondary breast lesions, (iii) across all breast lesions (iv) across axillary nodes (v) across supraclavicular nodes and (vi) across all nodes (vii) across all lesions (overall) using the following algorithm: CR: if measurement of '0' is noted at a given cycle as compared to baseline measurement which is >0 at screening or cycle 1 day 1; PR: if measurement is at least a 30% decreased compared to baseline levels . (Reference= baseline size or sum of sizes). Clinical Responders are participants who have achieved CR or PR during the Neo-adjuvant treatment. Overall response is derived based on the sum total of breast tumors and all nodes examined.
Time Frame: Baseline up to Cycle 4 (assessed at Baseline, Day 1 of Cycles 1-4 Pre-Surgery) Up to approximately 24 months
Population: ITT Population; Analysis was performed according to initial randomization. Number of participants analyzed = participants evaluable for this outcome and n = number participants analyzed in the specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 71 | 58 | 61 | 47
percentage of participants
  Primary Breast Tumor (n=71,58,61,47) | 67.6 [55.5 to 78.2] | 65.5 [51.9 to 77.5] | 49.2 [36.1 to 62.3] | 66.0 [50.7 to 79.1]
  Overall Response (n=71,53,55,43) | 67.6 [55.5 to 78.2] | 67.9 [53.7 to 80.1] | 47.3 [33.7 to 61.2] | 65.1 [49.1 to 79.0]

11. Secondary Outcome: Percentage of Participants Achieving Clinical Response During Neo-Adjuvant Period by Clinical Examination
Description: Tumor assessments were made based on the RECIST criteria - version 1.0 The clinical response at each cycle up to the last assessment prior to surgery was derived for: i) the primary breast lesion; (ii) across secondary breast lesions, (iii) across all breast lesions (iv) across axillary nodes (v) across supraclavicular nodes and (vi) across all nodes (vii) across all lesions (overall) using the following algorithm: CR: if measurement of '0' is noted at a given cycle as compared to baseline measurement which is >0 at screening or cycle 1 day 1; PR: if measurement is at least a 30% decreased compared to baseline levels . (Reference= baseline size or sum of sizes). Clinical Responders are participants who have achieved CR or PR during the Neo-adjuvant treatment. Primary breast tumor clinical response is based on primary breast tumor assessment. Overall response is derived based on the sum total of breast tumors and all nodes examined.
Time Frame: Baseline up to Cycle 4 (assessed at Baseline, Day 1 of Cycles 1-4 Pre-Surgery) Up to approximately 24 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 99 | 101 | 102 | 91
percentage of participants
  Primary Breast Tumor (n=99,101,102,91) | 79.8 [70.5 to 87.2] | 88.1 [80.2 to 93.7] | 67.6 [57.7 to 76.6] | 71.4 [61.0 to 80.4]
  Overall Response (n=97,100,98,88) | 81.4 [72.3 to 88.6] | 88.0 [80.0 to 93.6] | 66.3 [56.1 to 75.6] | 73.9 [63.4 to 82.7]

12. Secondary Outcome: Time to Clinical Response During Neo-Adjuvant Treatment Period
Description: Time to clinical response was defined as the time from the date of first dose received to the date of assessment of clinical response. Time to Clinical response was determined by Kaplan-Meier estimates. Tumor assessments were made based on the RECIST criteria - version 1.0. The clinical response at each cycle up to the last assessment prior to surgery was derived for: i) the primary breast lesion; (ii) across secondary breast lesions, (iii) across all breast lesions (iv) across axillary nodes (v) across supraclavicular nodes and (vi) across all nodes (vii) across all lesions (overall) using the following algorithm: CR: if measurement of '0' is noted at a given cycle as compared to baseline measurement which is >0 at screening or cycle 1 day 1; PR: if measurement is at least a 30% decreased compared to baseline levels . (Reference= baseline size or sum of sizes). Clinical Responders are participants who have achieved CR or PR during the Neo-adjuvant treatment.
Time Frame: Baseline up to Cycle 4 (assessed at Baseline, Day 1 of Cycles 1-4 Pre-Surgery) Up to approximately 24 months
Population: as for outcome 2
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 99 | 101 | 102 | 91
months | 6.3 [6.0 to 7.0] | 6.3 [4.0 to 7.0] | 6.9 [6.0 to 9.0] | 7.3 [6.0 to 9.0]

13. Secondary Outcome: Percentage of Participants With Progressive Disease During Neo-Adjuvant Treatment Period
Description: Tumor assessments were made based upon the Response Evaluation Criteria in Solid Tumors (RECIST) criteria - version 1.0. The clinical response at each cycle up to the last assessment prior to surgery was derived for: i) the primary breast lesion; (ii) across secondary breast lesions, (iii) across all breast lesions (iv) across axillary nodes (v) across supraclavicular nodes and (vi) across all nodes (vii) across all lesions (overall) using the following algorithm: PD: if lesion is at least a 20 % increased from measurements at baseline. Percentage of participants along with 95% Confidence Interval (CI) for one sample binomial using Pearson-Clopper method were reported. Missing investigator assessments were considered as no progressive disease.
Time Frame: Baseline up to Cycle 4 (assessed at Baseline, Day 1 of Cycles 1-4 Pre-Surgery) Up to approximately 24 months
Population: ITT Population; Analysis was performed according to initial randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Trastuzumab+Docetaxel: Neoadjuvant (Pre-Operative) Treatment: Participants received trastuzumab IV infusion at a loading dose of 8 mg/kg on Day 1 of Cycle 1 (21-day cycle) followed by a maintenance dose of 6 mg/kg on Day 1 of Cycles 2-4 and docetaxel IV infusion at a loading dose of 75 mg/m^2 on Day 1 of Cycle 1 followed by 100 mg/m^2 on Day 1 of Cycles 2-4, if no dose limiting toxicity occurred.
  Adjuvant (2-Week Post-Operative) Treatment: Participants received trastuzumab 6 mg/kg IV followed by FEC on Day 1 and every 3 weeks thereafter for three cycles (Cycles 5-7). Trastuzumab 6 mg/kg IV was continued every 3 weeks from Cycle 8 to Cycle 17.
- Trastuzumab+Pertuzumab+Docetaxel: Neoadjuvant (Pre-Operative) Treatment: Participants received trastuzumab IV infusion at a loading dose of 8 mg/kg and pertuzumab IV infusion at a loading dose of 840 mg on Day 1 of Cycle 1 (21-day cycle) followed by a maintenance dose of 6 mg/kg trastuzumab and 420 mg pertuzumab on Day 1 of Cycles 2-4. Docetaxel IV infusion was administered at a loading dose of 75 mg/m^2 on Day 1 of Cycle 1 followed by 100 mg/m^2 on Day 1 of Cycles 2-4, if no dose limiting toxicity occurred.
  Adjuvant (2-Week Post-Operative) Treatment: Participants received trastuzumab 6 mg/kg IV followed by FEC on Day 1 and every 3 weeks thereafter for three cycles (Cycles 5-7). Trastuzumab 6 mg/kg IV was continued every 3 weeks from Cycle 8 to Cycle 17.
- Pertuzumab+Docetaxel: Neoadjuvant (Pre-Operative) Treatment: Participants received pertuzumab IV at a loading dose of 840 mg on Day 1 of Cycle 1 (21-day cycle) followed by a maintenance dose of 420 mg on Day 1 of Cycles 2-4. Docetaxel IV infusion was administered at a loading dose of 75 mg/m^2 on Day 1 of Cycle 1 followed by 100 mg/m^2 on Day 1 of Cycles 2-4, if no dose limiting toxicity occurred.
  Adjuvant (2-Week Post-Operative) Treatment: Participants received trastuzumab 6 mg/kg IV followed by FEC on Day 1 and every 3 weeks thereafter for three cycles (Cycles 5-7). Trastuzumab 6 mg/kg IV was continued every 3 weeks from Cycle 8 to Cycle 21.
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 107 | 107 | 107 | 96
percentage of participants | 0.0 [0.0 to 3.4] | 0.9 [0.0 to 5.1] | 7.5 [3.3 to 14.2] | 2.1 [0.3 to 7.3]

14. Secondary Outcome: Percentage of Participants Achieving Breast Conserving Surgery For Whom Mastectomy Was Planned
Description: Breast Conserving Surgery (BCS) was defined as quadrantectomy, lumpectomy, no surgery, sentinel node biopsy, axillary surgical resection or other method of avoiding mastectomy.
Time Frame: Surgery (Within 2 weeks after Cycle 4) Up to approximately 24 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 62 | 56 | 61 | 60
percentage of participants | 22.6 [12.9 to 35.0] | 23.2 [13.0 to 36.4] | 18.0 [9.4 to 30.0] | 31.7 [20.3 to 45.0]

15. Secondary Outcome: Percentage of Participants Who Were Progression Free and Disease Free
Description: Disease-free survival (DFS) was defined as the time from first date of no disease to first documentation of PD or death. Participants without progression after surgery were considered Disease Free. Any evidence of contralateral disease in-situ was not considered as PD. Participants who were withdrawn from the study without documented progression and for whom evaluations were made, were censored at date of last assessment when participant was known to be disease-free. Progression-free survival (PFS) was defined as time from date of randomization to first documentation of PD or death. Any evidence of contralateral disease in-situ was not considered as PD. Participants who were withdrawn from study without documented progression and for whom evaluations were made, were censored at date of last assessment when the participant was known to be free from progressive disease. Participants without post baseline assessments but known to be alive were censored at the time of randomization.
Time Frame: Randomization up to a maximum of 329 weeks
Population: ITT Population; Analysis was performed according to initial randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 107 | 107 | 107 | 96
percentage of participants
  Progression Free | 82.2 | 84.1 | 74.8 | 75.0
  Disease Free | 82.5 | 85.1 | 80.2 | 76.1

16. Secondary Outcome: Progression Free and Disease Free Survival
Description: DFS was defined as the time from the first date of no disease (date of surgery) to the first documentation of PD or death. Participants without progression after surgery were considered Disease Free. Any evidence of contralateral disease in-situ was not considered as PD. PFS was defined as the time from the date of randomization to the first documentation of PD or death. Any evidence of contralateral disease in-situ was not considered as PD. DFS and PFS were determined using Kaplan-Meier estimates.
Time Frame: Randomization up to a maximum of 329 weeks
Population: ITT Population; Analysis was performed according to initial randomization.
Measure: Median (80% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Number analyzed (Participants) | 107 | 107 | 107 | 96
percentage of participants
  PFS | NA [NA to NA] — Median and corresponding 80% confidence interval were not achieved due to o the low number of events in this participant population, as expected. | 71.0 [71.0 to 76.0] | NA [NA to NA] — Median and corresponding 80% confidence interval were not achieved due to o the low number of events in this participant population, as expected. | NA [NA to NA] — Median and corresponding 80% confidence interval were not achieved due to o the low number of events in this participant population, as expected.
  DFS | NA [NA to NA] — Median and corresponding 80% confidence interval were not achieved due to o the low number of events in this participant population, as expected. | 67.2 [67.0 to 72.0] | NA [NA to NA] — Median and corresponding 80% confidence interval were not achieved due to o the low number of events in this participant population, as expected. | NA [NA to NA] — Median and corresponding 80% confidence interval were not achieved due to o the low number of events in this participant population, as expected.
Statistical Analysis 1: Comparison: Trastuzumab+Docetaxel vs Trastuzumab+Pertuzumab+Docetaxel; PFS; Test type: Superiority or Other; p = 0.2983, Cochran-Mantel-Haenszel; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.34 to 1.40] — HR is based on Cox proportional hazard regression stratified by breast cancer type and hormone positivity
Statistical Analysis 2: Comparison: Trastuzumab+Docetaxel vs Trastuzumab+Pertuzumab; PFS; Test type: Superiority or Other; p = 0.4722, Cochran-Mantel-Haenszel; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.68 to 2.30] — HR is based on Cox proportional hazard regression stratified by breast cancer type and hormone positivity
Statistical Analysis 3: Comparison: Trastuzumab+Pertuzumab+Docetaxel vs Pertuzumab+Docetaxel; PFS; Test type: Superiority or Other; p = 0.0268, Cochran-Mantel-Haenszel; Hazard Ratio (HR) = 2.05, 95% CI 2-sided [1.07 to 3.93] — HR is based on Cox proportional hazard regression stratified by breast cancer type and hormone positivity
Statistical Analysis 4: Comparison: Trastuzumab+Docetaxel vs Trastuzumab+Pertuzumab+Docetaxel; DFS; Test type: Superiority or Other; p = 0.1805, Cochran-Mantel-Haenszel; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.28 to 1.27] — HR is based on Cox proportional hazard regression stratified by breast cancer type and hormone positivity
Statistical Analysis 5: Comparison: Trastuzumab+Docetaxel vs Trastuzumab+Pertuzumab; DFS; Test type: Superiority or Other; p = 0.5901, Cochran-Mantel-Haenszel; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.42 to 1.64] — HR is based on Cox proportional hazard regression stratified by breast cancer type and hormone positivity
Statistical Analysis 6: Comparison: Trastuzumab+Pertuzumab+Docetaxel vs Pertuzumab+Docetaxel; DFS; Test type: Superiority or Other; p = 0.0250, Cochran-Mantel-Haenszel; Hazard Ratio (HR) = 2.16, 95% CI 2-sided [1.08 to 4.32] — HR is based on Cox proportional hazard regression stratified by breast cancer type and hormone positivity

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of Screening until the clinical cut off date 20th October 2014 up to 7 years.
Description: The safety population included all participants who received at least one dose of study medication and at least one safety assessment performed at baseline. Participants were assigned to treatment groups according to treatment actually received.
Arm/Group | Trastuzumab+Docetaxel | Trastuzumab+Pertuzumab+Docetaxel | Trastuzumab+Pertuzumab | Pertuzumab+Docetaxel
Serious Adverse Events (participants affected / at risk) | 21/107 | 22/107 | 19/108 | 21/94
Other Adverse Events (participants affected / at risk) | 107/107 | 105/107 | 101/108 | 94/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab+Docetaxel (N=107) | Trastuzumab+Pertuzumab+Docetaxel (N=107) | Trastuzumab+Pertuzumab (N=108) | Pertuzumab+Docetaxel (N=94)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 8 | 4 | 12
Neutropenia (Blood and lymphatic system disorders) | 1 | 6 | 3 | 6
Neutropenic infection (Infections and infestations) | 1 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 2 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 2 | 1
Imparied healing (General disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 3 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis fulminant (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dural arteriovenous fistula (Nervous system disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab+Docetaxel (N=107) | Trastuzumab+Pertuzumab+Docetaxel (N=107) | Trastuzumab+Pertuzumab (N=108) | Pertuzumab+Docetaxel (N=94)
Nausea (Gastrointestinal disorders) | 70 | 71 | 52 | 61
Diarrhoea (Gastrointestinal disorders) | 40 | 55 | 46 | 52
Vomiting (Gastrointestinal disorders) | 31 | 39 | 31 | 37
Stomatitis (Gastrointestinal disorders) | 12 | 22 | 21 | 11
Abdominal pain upper (Gastrointestinal disorders) | 8 | 9 | 12 | 12
Constipation (Gastrointestinal disorders) | 12 | 14 | 9 | 6
Abdominal pain (Gastrointestinal disorders) | 9 | 11 | 8 | 10
Haemorrhoids (Gastrointestinal disorders) | 5 | 8 | 8 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 6 | 6 | 5
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 75 | 73 | 59 | 65
Rash (Skin and subcutaneous tissue disorders) | 26 | 30 | 22 | 30
Nail disorder (Skin and subcutaneous tissue disorders) | 17 | 13 | 16 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5 | 10 | 8
Erythema (Skin and subcutaneous tissue disorders) | 5 | 6 | 7 | 11
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 7 | 2 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 6 | 4 | 7
Acne (Skin and subcutaneous tissue disorders) | 3 | 7 | 2 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 2 | 3 | 2
Fatigue (General disorders) | 35 | 35 | 34 | 37
Mucosal inflammation (General disorders) | 28 | 33 | 18 | 28
Asthenia (General disorders) | 22 | 29 | 19 | 23
Pyrexia (General disorders) | 16 | 25 | 21 | 14
Oedema peripheral (General disorders) | 12 | 7 | 18 | 9
Chills (General disorders) | 8 | 4 | 10 | 2
Chest pain (General disorders) | 4 | 2 | 4 | 6
Pain (General disorders) | 2 | 3 | 3 | 7
Oedema (General disorders) | 1 | 0 | 6 | 4
Neutropenia (Blood and lymphatic system disorders) | 80 | 64 | 46 | 67
Leukopenia (Blood and lymphatic system disorders) | 24 | 13 | 13 | 15
Anaemia (Blood and lymphatic system disorders) | 9 | 6 | 11 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 25 | 29 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 18 | 13 | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 13 | 5 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 11 | 7 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 8 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7 | 7 | 6
Headache (Nervous system disorders) | 17 | 14 | 25 | 22
Dysgeusia (Nervous system disorders) | 16 | 16 | 14 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 10 | 15 | 14
Dizziness (Nervous system disorders) | 8 | 6 | 14 | 8
Neuropathy peripheral (Nervous system disorders) | 10 | 6 | 4 | 5
Paraesthesia (Nervous system disorders) | 7 | 2 | 3 | 5
Radiation skin injury (Injury, poisoning and procedural complications) | 21 | 19 | 22 | 24
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 7 | 8 | 8
Seroma (Injury, poisoning and procedural complications) | 6 | 7 | 4 | 5
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3 | 6 | 2
Incision site pain (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 19 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 11 | 6 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 2 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 12 | 9 | 11 | 13
Nasopharyngitis (Infections and infestations) | 12 | 8 | 7 | 5
Pharyngitis (Infections and infestations) | 8 | 4 | 4 | 5
Urinary tract infection (Infections and infestations) | 7 | 4 | 3 | 6
Hot flush (Vascular disorders) | 11 | 12 | 8 | 7
Lymphoedema (Vascular disorders) | 4 | 6 | 12 | 5
Flushing (Vascular disorders) | 6 | 5 | 5 | 5
Hypertension (Vascular disorders) | 5 | 6 | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 19 | 18 | 15 | 23
Insomnia (Psychiatric disorders) | 14 | 13 | 8 | 14
Anxiety (Psychiatric disorders) | 2 | 3 | 6 | 0
Alanine aminotransferase increased (Investigations) | 9 | 2 | 2 | 5
Weight increased (Investigations) | 4 | 2 | 9 | 1
Aspartate aminotransferase increased (Investigations) | 9 | 0 | 2 | 2
Palpitations (Cardiac disorders) | 2 | 5 | 7 | 5
Left ventricular dysfunction (Cardiac disorders) | 2 | 6 | 2 | 5
Menstruation irregular (Reproductive system and breast disorders) | 7 | 4 | 10 | 9
Drug hypersensitivity (Immune system disorders) | 2 | 6 | 12 | 6
Lacrimation increased (Eye disorders) | 3 | 8 | 6 | 6
General Disorder (General disorders) | 17 | 16 | 15 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.